CLINICAL TRIAL: NCT05874713
Title: A Phase 2, Multi-Center, Randomized, Observer-Blind Study, to Evaluate Safety and Immunogenicity of Homologous or Heterologous Priming and Booster Vaccinations With H5N8 or H5N6 MF59-adjuvanted, Cell Culture-derived Influenza Vaccine in Healthy Subjects ≥18 Years of Age
Brief Title: Study to Evaluate Safety and Immunogenicity of Different Priming and Booster Regimens With Adjuvanted H5N8 and/or H5N6 Influenza Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V205_01
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Influenza, Human; Infections; Respiratory Tract Infections; Virus Diseases; Infection Viral
Keywords: Influenza; Vaccine; MF59; Adjuvant; H5N8; H5N6; Pandemic; Avian
MeSH Terms: conditions — Influenza, Human; Infections; Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Eligible subjects are randomized in a 2:1:1 ratio to Treatment Arm A, B, or C, respectively, and will receive two priming doses of the allocated aH5N8c/aH5N6c vaccine 3 weeks apart, ie, at Day 1 and Day 22, and a booster dose of aH5N8c vaccine at Day 202.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Eligible subjects who have been randomized to receive aH5N8c on Day 1, Day 22 and Day 202
  Interventions: Biological: aH5N8c on Day 1; Biological: aH5N8c on Day 22; Biological: aH5N8c on Day 202
- Arm B (Experimental): Eligible subjects who have been randomized to receive aH5N8c on Day 1, aH5N6c on Day 22, and aH5N8c on Day 202
  Interventions: Biological: aH5N8c on Day 1; Biological: aH5N6c on Day 22; Biological: aH5N8c on Day 202
- Arm C (Experimental): Eligible subjects who have been randomized to receive aH5N6c on Day 1 and aH5N8c on Day 22 and Day 202
  Interventions: Biological: aH5N6c on Day 1; Biological: aH5N8c on Day 22; Biological: aH5N8c on Day 202

INTERVENTIONS:
Biological: aH5N8c on Day 1 — MF59-adjuvanted cell-culture derived subunit inactivated monovalent A/H5N8 vaccine (aH5N8c) for intramuscular administration, containing intermediate dose H5N8 hemagglutinin + standard dose MF59 (approximately 0.5 mL total volume)
  Arms: Arm A; Arm B
Biological: aH5N6c on Day 1 — MF59-adjuvanted cell-culture derived subunit inactivated monovalent A/H5N6 vaccine (aH5N6c) for intramuscular administration, containing intermediate dose H5N6 hemagglutinin + standard dose MF59 (approximately 0.5 mL total volume)
  Arms: Arm C
Biological: aH5N8c on Day 22 — MF59-adjuvanted cell-culture derived subunit inactivated monovalent A/H5N8 vaccine (aH5N8c) for intramuscular administration, containing intermediate dose H5N8 hemagglutinin + standard dose MF59 (approximately 0.5 mL total volume)
  Arms: Arm A; Arm C
Biological: aH5N6c on Day 22 — MF59-adjuvanted cell-culture derived subunit inactivated monovalent A/H5N6 vaccine (aH5N6c) for intramuscular administration, containing intermediate dose H5N6 hemagglutinin + standard dose MF59 (approximately 0.5 mL total volume)
  Arms: Arm B
Biological: aH5N8c on Day 202 — MF59-adjuvanted cell-culture derived subunit inactivated monovalent A/H5N8 vaccine (aH5N8c) for intramuscular administration, containing intermediate dose H5N8 hemagglutinin + standard dose MF59 (approximately 0.5 mL total volume)

SUMMARY:
This Phase 2, randomized, observer-blind clinical study is evaluating 3 different priming and booster regimens with MF59-adjuvanted H5N8 and/or H5N6 cell culture-derived influenza vaccine (aH5N8c; aH5N6c). Approximately 480 healthy adult subjects are to be randomized into 1 of 3 possible treatment groups, stratified by age group (18-64 years and ≥65 years) and by poultry worker status (yes/no). Each subject will receive a priming influenza vaccine injection on Day 1 and Day 22 and a booster vaccination on Day 202. Subjects will be followed up for approximately 6 months after the booster injection.

The primary immunogenicity analysis is based on antibody responses against H5N8 and H5N6 as measured by hemagglutination inhibition (HI) assay on Day 1, Day 22, Day 29, Day 43, Day 202, Day 209 (H5N8 only), and Day 223.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of ≥18 years of age on the day of informed consent.
* Individuals who or whose legally acceptable representative(s) have voluntarily given written consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
* Individuals who can comply with study procedures including follow-up.
* Males, females of non-childbearing potential or females of childbearing potential who are using an effective birth control method which they intend to use for at least 30 days before the first study vaccination and plan to do so until 2 months after the last study vaccination.
* Individuals must provide a baseline blood sample prior to randomization and vaccination.

Exclusion Criteria:

* Females of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of contraceptive methods from at least 30 days prior to study entry and who do not plan to do so until 2 months after the last study vaccination.
* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Abnormal function of the immune system resulting from:

  1. Clinical conditions.
  2. Systemic administration of corticosteroids at a dose ≥20 mg/day of prednisone (or equivalent) for more than 14 consecutive days within 90 days prior to informed consent. Topical, inhaled and intranasal corticosteroids are permitted. Intermittent use (one dose in 30 days) of intra-articular corticosteroids are also permitted.
  3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
* History of any medical condition considered an AESI.
* Received immunoglobulins with immunomodulating effects or any blood products within 180 days prior to informed consent.
* Individuals who previously received an H5 influenza vaccine or have a known history of H5 influenza infection prior to enrollment.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent or are unwilling to refuse participation in another clinical study at any time during the conduct of this study.
* Study personnel or immediate family or household member of study personnel.
* Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the individual due to participation in the study.
* Individuals who received any other vaccines (with the exception of COVID-19 vaccines) within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from any of the 3 scheduled study vaccinations.
* Receipt of any (investigational or licensed) COVID-19 vaccine within 14 days (non-replicating vaccines) or 28 days (replicating vaccines) prior to enrollment or plan to receive any COVID-19 vaccine within 7 days from any of the 3 scheduled study vaccinations.
* A known history of Guillain-Barre Syndrome or other demyelinating diseases such as encephalomyelitis and transverse myelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of hemagglutination inhibition (HI) antibodies against H5N8 strain - Day 1 | Day 1
  GMT (HI) prevaccination
GMT of HI antibodies against H5N8 strain - Day 22 | Day 22
  GMT (HI) 3 weeks post first priming vaccination
GMT of HI antibodies against H5N8 strain - Day 43 | Day 43
  GMT (HI) 3 weeks post second priming vaccination
GMT of HI antibodies against H5N8 strain - Day 202 | Day 202
  GMT (HI) pre booster vaccination
GMT of HI antibodies against H5N8 strain - Day 209 | Day 209
  GMT (HI) 1 week post booster vaccination
GMT of HI antibodies against H5N8 strain - Day 223 | Day 223
  GMT (HI) 3 weeks post booster vaccination
GMT of HI antibodies against H5N6 strain - Day 1 | Day 1
  GMT (HI) prevaccination
GMT of HI antibodies against H5N6 strain - Day 22 | Day 22
  GMT (HI) 3 weeks post first priming vaccination
GMT of HI antibodies against H5N6 strain - Day 43 | Day 43
  GMT (HI) 3 weeks post second priming vaccination
GMT of HI antibodies against H5N6 strain - Day 202 | Day 202
  GMT (HI) pre booster vaccination
GMT of HI antibodies against H5N6 strain - Day 223 | Day 223
  GMT (HI) 3 weeks post booster vaccination
Geometric mean fold increase (GMFI) of HI antibodies against H5N8 strain - Day 22 | Day 22
  GMFI (HI) 3 weeks post first priming vaccination compared to prevaccination
GMFI of HI antibodies against H5N8 strain - Day 43 | Day 43
  GMFI (HI) 3 weeks post second priming vaccination compared to prevaccination
GMFI of HI antibodies against H5N8 strain - Day 209 | Day 209
  GMFI (HI) 1 week post booster vaccination compared to pre booster vaccination
GMFI of HI antibodies against H5N8 strain - Day 223 | Day 223
  GMFI (HI) 3 weeks post booster vaccination compared to pre booster vaccination
GMFI of HI antibodies against H5N6 strain - Day 22 | Day 22
  GMFI (HI) 3 weeks post first priming vaccination compared to prevaccination
GMFI of HI antibodies against H5N6 strain - Day 43 | Day 43
  GMFI (HI) 3 weeks post second priming vaccination compared to prevaccination
GMFI of HI antibodies against H5N6 strain - Day 223 | Day 223
  GMFI (HI) 3 weeks post booster vaccination compared to pre booster vaccination
Percentages of subjects with HI titers ≥1:40 against H5N8 strain - Day 1 | Day 1
  % ≥1:40 (HI) prevaccination
Percentages of subjects with HI titers ≥1:40 against H5N8 strain - Day 22 | Day 22
  % ≥1:40 (HI) 3 weeks post first priming vaccination
Percentages of subjects with HI titers ≥1:40 against H5N8 strain - Day 43 | Day 43
  % ≥1:40 (HI) 3 weeks post second priming vaccination
Percentages of subjects with HI titers ≥1:40 against H5N8 strain - Day 209 | Day 209
  % ≥1:40 (HI) 1 week post booster vaccination
Percentages of subjects with HI titers ≥1:40 against H5N8 strain - Day 223 | Day 223
  % ≥1:40 (HI) 3 weeks post booster vaccination
Percentages of subjects with HI titers ≥1:40 against H5N6 strain - Day 1 | Day 1
  % ≥1:40 (HI) prevaccination
Percentages of subjects with HI titers ≥1:40 against H5N6 strain - Day 22 | Day 22
  % ≥1:40 (HI) 3 weeks post first priming vaccination
Percentages of subjects with HI titers ≥1:40 against H5N6 strain - Day 43 | Day 43
  % ≥1:40 (HI) 3 weeks post second priming vaccination
Percentages of subjects with HI titers ≥1:40 against H5N6 strain - Day 223 | Day 223
  % ≥1:40 (HI) 3 weeks post booster vaccination
Percentages of subjects with seroconversion by HI against H5N8 strain - Day 22 | Day 22
  % seroconversion (HI) 3 weeks post first priming vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with prevaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
Percentages of subjects with seroconversion by HI against H5N8 strain - Day 43 | Day 43
  % seroconversion (HI) 3 weeks post second priming vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
Percentages of subjects with seroconversion by HI against H5N8 strain - Day 209 | Day 209
  % seroconversion (HI) 1 week post booster vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
Percentages of subjects with seroconversion by HI against H5N8 strain - Day 223 | Day 223
  % seroconversion (HI) 3 weeks post booster vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
Percentages of subjects with seroconversion by HI against H5N6 strain - Day 22 | Day 22
  % seroconversion (HI) 3 weeks post first priming vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
Percentages of subjects with seroconversion by HI against H5N6 strain - Day 43 | Day 43
  % seroconversion (HI) 3 weeks post second priming vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
Percentages of subjects with seroconversion by HI against H5N6 strain - Day 223 | Day 223
  % seroconversion (HI) 3 weeks post booster vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10

SECONDARY OUTCOMES:
Frequency and severity of solicited local and systemic adverse events (AEs) | Day 1 through Day 7, Day 22 through Day 28, and Day 202 through 208
  For 7 consecutive days following each vaccination (ie, Day 1 through Day 7, Day 22 through Day 28, and Day 202 through 208, or until symptom resolution if ongoing at Day 7, Day 28 or Day 208 for a maximum of 14 days postvaccination).
Frequency and severity of unsolicited AEs | Day 1 through Day 43 and Day 202 through Day 223
  For 3 weeks following each vaccination
Frequency and severity of serious AEs (SAEs), AEs leading to withdrawal, AEs of special interest (AESI), and medically attended AEs (MAAEs) | Day 1 through Day 382
  From first vaccination until study completion
GMT of HI antibodies against H5N8 strain - Persistence | Day 202, Day 382
  GMT (HI) 6 months post 2nd priming vaccination and 6 months post booster vaccination
GMT of HI antibodies against H5N6 strain - Persistence | Day 202
  GMT (HI) 6 months post 2nd priming vaccination
GMFI of HI antibodies against H5N8 strain - Persistence | Day 202, Day 382
  GMFI (HI) 6 months post 2nd priming vaccination compared to prevaccination (Day 1), and 6 months post booster vaccination compared to prevaccination (Day 1) and compared to pre booster vaccination (Day 202)
GMFI of HI antibodies against H5N6 strain - Persistence | Day 202
  GMFI (HI) 6 months post 2nd priming vaccination compared to prevaccination
Percentages of subjects with HI titers ≥1:40 against H5N8 strain - Persistence | Day 202, Day 382
  % ≥1:40 (HI) 6 months post 2nd priming vaccination and 6 months post booster vaccination
Percentages of subjects with HI titers ≥1:40 against H5N6 strain - Persistence | Day 202
  % ≥1:40 (HI) 6 months post 2nd priming vaccination
Percentages of subjects with seroconversion by HI against H5N8 strain - Persistence | Day 202, Day 382
  % seroconversion (HI) 6 months post 2nd priming vaccination and 6 months post booster vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
Percentages of subjects with seroconversion by HI against H5N6 strain - Persistence | Day 202
  % seroconversion (HI) 6 months post 2nd priming vaccination, defined as a ≥4-fold increase in HI titer postvaccination in those with pre-vaccination titer ≥1:10, or a postvaccination HI titer ≥1:40 for subjects with prevaccination titer <1:10
GMT of microneutralization (MN) antibodies against H5N8 strain | Day 1, Day 22, Day 43, Day 202, Day 223
  GMT (MN) prevaccination, 3 weeks post priming vaccinations, pre booster vaccination and 3 weeks post booster vaccination
GMT of MN antibodies against H5N6 strain | Day 1, Day 43, Day 202, Day 223
  GMT (MN) prevaccination, 3 weeks post 2nd priming vaccination, pre booster vaccination and 3 weeks post booster vaccination
GMFI of MN antibodies against H5N8 strain | Day 22, Day 43, Day 202, Day 223
  GMFI (MN) 3 weeks post priming vaccinations and 6 months post 2nd priming vaccination compared to prevaccination (Day 1), and 3 weeks post booster vaccination compared to pre booster vaccination (Day 202)
GMFI of MN antibodies against H5N6 strain | Day 43, Day 202, Day 223
  GMFI (MN) 3 weeks and 6 months post 2nd priming vaccination compared to prevaccination (Day 1), and 3 weeks post booster vaccination compared to pre booster vaccination (Day 202)
Percentages of subjects with MN titers ≥1:40 against H5N8 strain | Day 1, Day 22, Day 43, Day 202, Day 223
  % ≥1:40 (MN) prevaccination, 3 weeks post priming vaccinations, pre booster vaccination, and 3 weeks post booster vaccination
Percentages of subjects with MN titers ≥1:40 against H5N6 strain | Day 1, Day 43, Day 202, Day 223
  % ≥1:40 (MN) prevaccination, 3 weeks post 2nd priming vaccination, pre booster vaccination, and 3 weeks post booster vaccination
Percentages of subjects with seroconversion by MN against H5N8 strain | Day 22, Day 43, Day 202, Day 209, Day 223
  % seroconversion (MN) 3 weeks post priming vaccinations, pre booster vaccination, and 3 weeks post booster vaccination, defined as a ≥4-fold increase in MN titer postvaccination for subjects with prevaccination titer ≥lower limit of quantification (LLOQ), or a postvaccination MN titer ≥4×LLOQ for subjects with prevaccination titer <LLOQ
Percentages of subjects with seroconversion by MN against H5N6 strain | Day 43, Day 202, Day 209, Day 223
  % seroconversion (MN) 3 weeks post 2nd priming vaccination, pre booster vaccination, and 3 weeks post booster vaccination, defined as a ≥4-fold increase in MN titer postvaccination for subjects with prevaccination titer ≥lower limit of quantification (LLOQ), or a postvaccination MN titer ≥4×LLOQ for subjects with prevaccination titer <LLOQ

CONTACTS AND LOCATIONS:
Overall Officials: Therapeutic Area Head, Study Chair — Seqirus
Locations (9):
- United States (9):
  - Cullman Clinical Trials, Cullman, Alabama
  - Lifeline Primary Care, Lilburn, Georgia
  - Georgia Clinic, Norcross, Georgia
  - Velocity Clinical Research, Sioux City, Iowa
  - Velocity Clinical Research, Baton Rouge, Louisiana
  - Velocity Clinical Research, Grand Island, Nebraska
  - Velocity Clinical Research, Norfolk, Nebraska
  - Medical Care LLC, Elizabethton, Tennessee
  - Cope Family Medicine, Bountiful, Utah

IPD SHARING:
Plan to Share IPD: Undecided